CLINICAL TRIAL: NCT03733938
Title: Outcome of Periradicular Microsurgery Using a Bioceramic Root End Filling Material
Brief Title: Microsurgery Using a Bioceramic Root End Filling Material
Acronym: microsurgery
Status: Completed | Type: Observational
Sponsor: Jordan University of Science and Technology (Other)
Responsible Party: Sponsor
Other Study IDs: 316/2016
Record Dates: First submitted 2018-11-05; First posted 2018-11-07 (Actual); Last update posted 2018-11-07 (Actual); Status verified 2018-11

CONDITIONS: Bone Resorption; Symptoms
Keywords: rarifaction; root end filling; bioceramic; outcome
MeSH Terms: conditions — Bone Resorption

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- teeth with failed root canal treatement: endodontic microsurgery will be performed for teeth with failed root canal treatment
  Interventions: Other: endodontic microsurgery

INTERVENTIONS:
Other: endodontic microsurgery — teeth with failed root canal treatment will be treated by endodontic microsurgery

SUMMARY:
Endodontic failures are not uncommonly encountered despite improvements in routine root canal therapy. Endodontic microsurgery is one way to manage such failure. The placement of a retrograde filling material is considered the most important prognostic factor in endodontic microsurgery. The aim of this study was to investigate the clinical and radiographic outcome of a fast set bioceramic root end filling material in human teeth.

DETAILED DESCRIPTION:
Patients who were referred to the endodontic postgraduate clinics in the period between January 2017 till August 2017 were assessed for inclusion in the study according to preset criteria. Endodontic microsurgery was performed following modern techniques including magnification, root resection with minimal angle, ultrasonic root end preparation and placement of a fast set bioceramic putty as retrograde filling material. The case was subsequently evaluated clinically and radiographically at 3, 6 and 12 months. And will be followed subsequently at 2 years and 4 years post treatment.

ELIGIBILITY:
Inclusion Criteria:

1. medically fit patient
2. Tooth has adequate coronal seala nd judged restorable
3. previously root filled tooth with persistent periapical lesion
4. previously retreated tooth with persistent symptoms 5.previously tretaed tooth with inaccessable canal for retreatment 6. combined nonsurgical and surgical approach for teeth with large periapical lesions

Exclusion Criteria:

* medically compromised patients
* nonrestorable teeth cracked roots

Ages: 16 Years to 70 Years | Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: All eligible patients attending the postgraduate clinics over a 7 months period and meet the inclusion criteria will be included in the study
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2017-01-06 (Actual); Primary Completion 2017-08-07 (Actual); Study Completion 2018-08-05 (Actual)

PRIMARY OUTCOMES:
Resolution of signs of failure in the root treated tooth | 6 months -1 year
  symptoms should disappear and signs of bone healing should be evident on the radio graph

CONTACTS AND LOCATIONS:
Overall Officials: Nessrin Taha, DCD, Study Chair — Jordan University of Science and Technology
Locations (1):
- Dental teaching centre, Irbid, Jordan

IPD SHARING:
Plan to Share IPD: Undecided
participant data can be shared after the first publication from the study.

REFERENCES:
- [Derived] Taha NA, Aboyounes FB, Tamimi ZZ. Root-end microsurgery using a premixed tricalcium silicate putty as root-end filling material: a prospective study. Clin Oral Investig. 2021 Jan;25(1):311-317. doi: 10.1007/s00784-020-03365-7. Epub 2020 Jun 2. PMID 32483680